CLINICAL TRIAL: NCT05352659
Title: Increasing Effective Mental Health Care for LGBT Clients
Acronym: UMD-PRC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Brad Boekeloo, Professor, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: U48DP006382 (NIH)
Record Dates: First submitted 2021-12-16; First posted 2022-04-29 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Sexual Orientation; Gender Identity
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Provider skills assessors will be masked to condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face and online LGBTQ training+ (Experimental): The Study Intervention arm receives the organization-level LGBTQ climate assessment and technical assistance, the provider-level face-to-face LGBTQ training along with links to publicly available on-line training.
  Interventions: Behavioral: Face-to-face and online LGBTQ+ training
- On-line resources (Other): The Comparison Intervention arm receives only links to publicly available on-line resources.
  Interventions: Behavioral: On-line training

INTERVENTIONS:
Behavioral: Face-to-face and online LGBTQ+ training — The intervention consists of Organization-level technical assistance in regard to LGBTQ climate of the organization AND Clinician-level face-to-face virtual workshop LGBTQ competency training, virtual clinical consultations, and links to publicly available LGBTQ training.
  Arms: Face-to-face and online LGBTQ training+
Behavioral: On-line training — This study arm receives only links to publicly available on-line LGBTQ training.
  Arms: On-line resources

SUMMARY:
The overall aims of the 5-year University of Maryland Prevention Research Center (UMD-PRC) Core Research Project are to identify, refine, implement, evaluate, translate, disseminate, and communicate approaches and tools that can be used to improve the competency of mental health care for LGBT persons which is a social determinant of LGBT health disparities. The UMD-PRC research team, in collaboration with the community advisory board (CAB), have identified 5 evidence based resources (Tools) to improve health care competency with sexual and gender minority populations (lesbian/gay, bisexual, and transgender [LGBT] people). The UMD-PRC will use the Sexual and Gender Diversity Learning Community (SGDLC) program (Strategy) and these tools along with technical assistance (TA) to improve LGBT mental health care. The following hypothesis will be tested. The study intervention group will show an increase in a) organization-level LGBT-friendly policies and environment as observed by the researchers and b) LGBT competent clinician practice assessed through clinician self-reported preparedness, awareness, and knowledge as well as referral for co-occurring client health needs; client-reported satisfaction with therapy and health literacy; and research team assessment of clinician performance providing consultation to a standardized LGBT patient actor.

DETAILED DESCRIPTION:
Mental health organizations will be randomized to two study groups. Within each organization, clinicians will be recruited. Within clinician practices, clients will be recruited. Baseline data will be collected from the two groups of mental health organization leads, clinicians, and clients. Both groups will undergo data collection with 5 tools by research teams: at the organization level the Organizational Climate Assessment and at the clinician level the Provide Self-Assessment during month 1 of each site's participation. Client level Client Satisfaction Survey data will also be collected during month 1 of each site's participation (cohort 1 clients). During months 2-4 of each site's participation, clinicians in the control group will receive standard nationally, publicly freely accessible information, specifically a letter notifying them about the on-line accessible SAMHSA LGBT services education manual and Fenway Health Webinars. In the intervention group, clinicians will also receive a letter notifying them about the nationally, publicly freely accessible on-line SAMHSA education manual and Fenway Health Webinars plus they will receive a 1-day, clinician training followed by 4 biweekly 2-hour technical assistance workshops to review and address information gleaned from the 5 tool's and to finalize the problem-solving related to needs for change based on the 5 tool's. During month 5 of each site's participation, both groups will undergo follow-up data collection and assessment by research teams at the organization and clinician levels. Client level data will also be collected during month 5 of each site's participation (cohort 2 clients). Finally, during month 6 of each site's participation, each site's 5 clinicians in both study arms will complete one first-time consultation session by screen-to-screen interaction via on-line computer interface with a LGBT standardized patient so that their objective skill-level performance can be assessed.

ELIGIBILITY:
Inclusion Criteria:

Therapists must be employed by a participating study general mental health services organization in Maryland. They must be 18 years of age or older, in the process of being licensed or already licensed to provide clinical mental healthcare in Maryland, able to speak and understand English, and have at least 10 clients 16 years old and older.

Exclusion Criteria:

Participants may not be under 18 years of age, unlicensed, or have less than 10 clients 16 years or older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Virtual Simulated Client Skill Assessment | Within 30 days after therapist completion of the intervention, an average of 6 months after enrollment.
  Therapists' conduct an initial consultation visit through an on-line interface with an actor trained to follow a specific client LGBTQ profile and the therapists' skills with the simulated client are assessed using a standardized performance checklist by researchers while they view an audio-video recording of the visit.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Boekeloo, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland School of Public Health, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Under appropriate circumstances the investigators will share de-identified client-level data with other qualified investigators.

DOCUMENTS (1):
  • Informed Consent Form (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT05352659/ICF_000.pdf